CLINICAL TRIAL: NCT07114692
Title: The Effect of Intradermal Stromal Vascular Fraction Transplantation on the Regeneration of Expanded Skin: a Randomized Controlled Trial
Brief Title: The Effect of Stromal Vascular Fraction Transplantation on the Regeneration of Expanded Skin
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Tao Zan, MD, Ph.D, Vice Director of the Department of Plastic and Reconstructive Surgery, Shanghai Ninth People's Hospital, SJTUSM, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shanghai9th-SVF-ES-RCT
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-06

CONDITIONS: Skin Regeneration
Keywords: skin expansion; stromal vascular fraction
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stromal vascular fraction transplantation (Experimental): Subcutaneous fat was harvested from either the abdomen or the posterior inner thigh region and then digested with 600 U of collagenase (Shanghai Qiaoyuan Biological Pharmaceutical Co., Ltd, Shanghai, China) at 37°C and 150rpm for three hours. After enzymatic digestion, the lower aqueous phase liquid was aspirated to acquire the stromal vascular fraction (SVF). The SVF cell-pellet was washed and adjusted to 2×10^6 cells/mL. Lidocaine cream will be applied to the expanded skin to achieve surface anesthesia. The skin was marked with methylene blue and a total of 0.5ml (around 1×10^6 cells) were transplanted intradermally at the center of each 2cm×2cm squares. The expander was inflated two times a week using constant pressure inflation method, where the intracapsular pressure was monitored using a pressure meter and the inflation was halted when the pressure reached 100 mmHg.
  Interventions: Biological: Stromal vascular fraction transplantation
- Normal saline injection (Placebo Comparator): Lidocaine cream will be applied to the expanded skin to achieve surface anesthesia. The skin was marked with methylene blue and a total of 0.5ml 0.9% normal saline were transplanted intradermally at the center of each 2cm×2cm squares. The expander was inflated two times a week using constant pressure inflation method, where the intracapsular pressure was monitored using a pressure meter and the inflation was halted when the pressure reached 100 mmHg.
  Interventions: Biological: Normal saline injection

INTERVENTIONS:
Biological: Stromal vascular fraction transplantation — Subcutaneous fat was harvested from either the abdomen or the posterior inner thigh region and then digested with 600 U of collagenase (Shanghai Qiaoyuan Biological Pharmaceutical Co., Ltd, Shanghai, China) at 37°C and 150rpm for three hours. After enzymatic digestion, the lower aqueous phase liquid was aspirated to acquire the stromal vascular fraction (SVF). The SVF cell-pellet was washed and adjusted to 2×10^6 cells/mL. Lidocaine cream will be applied to the expanded skin to achieve surface anesthesia. The skin was marked with methylene blue and a total of 0.5ml (around 1×10^6 cells) were transplanted intradermally at the center of each 2cm×2cm squares. The expander was inflated two times a week using constant pressure inflation method, where the intracapsular pressure was monitored using a pressure meter and the inflation was halted when the pressure reached 100 mmHg.
  Arms: Stromal vascular fraction transplantation
Biological: Normal saline injection — Lidocaine cream will be applied to the expanded skin to achieve surface anesthesia. The skin was marked with methylene blue and a total of 0.5ml 0.9% normal saline were transplanted intradermally at the center of each 2cm×2cm squares. The expander was inflated two times a week using constant pressure inflation method, where the intracapsular pressure was monitored using a pressure meter and the inflation was halted when the pressure reached 100 mmHg.
  Arms: Normal saline injection

SUMMARY:
This study is a randomized controlled trial aimed at evaluating the effect of intradermal stromal vascular fraction (SVF) transplantation in treating exhaustion of dermal regenerative capacity during skin expansion. The dermal thickness, texture, and perfusion before and after SVF transplantation would be recorded and analyzed by a series of quantitative devices including laser 3D scanner, ultrasound, VISIA skin analyzer, CK skin analyzer, and indocyanine green angiography.

DETAILED DESCRIPTION:
This study is a randomized controlled trial aimed at evaluating the effect of intradermal stromal vascular fraction (SVF) transplantation in treating exhaustion of dermal regenerative capacity during skin expansion. This study will enroll patients experiencing dermal exhaustion during the process of skin soft tissue expansion. Participants will be randomly assigned in a 1:1 ratio to either the stromal vascular fraction (SVF) transplantation group or the normal saline control group. To confirm eligibility, all potential participants will undergo a baseline screening visit. Those meeting the inclusion criteria will proceed to the study center for enrollment assessment, followed by randomization. Participants in the SVF transplantation group will undergo abdominal liposuction and receive intradermal SVF transplantation. Participants in the control group will receive intradermal injections of an equivalent volume of normal saline. The changes of dermis of expanded skin were recorded before the treatment (baseline), and at 4 weeks and 8 weeks follow-up timepoints after SVF transplantation. More specifically, skin surface area was measured using laser 3D scan; skin thickness and texture were detected by ultrasound, VISIA skin analyzer and CK skin analyzer; skin blood perfusion was analyzed using indocyanine green angiography.

ELIGIBILITY:
Inclusion Criteria:

* Age: over 18 years and under 65 years;
* show signs of deterioration of skin texture during expansion, including stretch marks or thinning of the dermis;
* Have signed the informed consent form, agree to participate in this study, and are able to comply with follow-up requirements.

Exclusion Criteria:

* Patients with serious underlying diseases such as cardiovascular or cerebrovascular disease, peripheral vascular disease, or impaired liver or kidney function;
* Patients with a long history of smoking and alcohol use who have not quit smoking or drinking;
* Patients allergic to iodine or iodine-containing preparations;
* Patients with psychiatric disorders, lack of insight, or those who cannot accurately express themselves or cooperate;
* Patients with contraindications for SVF transplantation, such as ulceration or infection of the expanded skin;
* Patients with severely loose skin or insufficient subcutaneous fat tissue;
* Patients who request to withdraw informed consent and exit the clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Dermal thickness | Baseline, 4 and 8 weeks after intervention
  Using Doppler ultrasound to measure the full-thickness of skin dermis of the expanded skin. The measurements were conducted at the center of the expanded skin and other four points (above, below, left, right) around the center. The average value is taken to represent the dermal thickness of the patient's expanded skin.

SECONDARY OUTCOMES:
Skin surface area | baseline, 4 and 8 weeks after intervention
  Using the HSCAN771 handheld laser 3D scanner and the VIVID910 3D laser scanning system to measure the surface area of the expanded skin.

OTHER OUTCOMES:
Skin texture | Baseline, 4 and 8 weeks after intervention
  Using the VISIA skin analyzer to visualize the distribution of dermal marks, which is an indication of dermal rupture. Briefly, photographs of the patient's expanded skin were taken from three standard angles: front, left side, and right side. Use the VISIA instrument to generate texture imaging of the expanded skin, selecting the expanded skin and surrounding normal skin as the region of interest. Employ the instrument's built-in red area analysis function to analyze the distribution of dermal marks in the expanded skin.
  Using the elasticity probe of CK Skin analyzer to measure the elasticity of the expanded skin. Represent skin softness through the skin viscoelasticity parameter R2 (R2 = Ua/Uf, where Ua is the total elastic and plastic recovery, and Uf is the total elastic and plastic deformation).
Skin perfusion | Baseline, 4 and 8 weeks after intervention
  Indocyanine green (ICG) angiography was used to detect the blood perfusion of the expanded skin. Briefly, the detector of SPY imaging system was adjusted to approximately 20 cm from the surface of the flap. A white light photograph of the expanded skin was taken. Without changing the detector position, indocyanine green imaging was performed as follows: Inject 2 ml of ICG solution (2.5 mg/ml) intravenously and fluorescence signals from the expanded skin were collected by SPY imaging system. The integrated SPY-Q software was used for the analysis of the arterial and venous perfusion of the expanded flap.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zan, M.D., Ph.D., Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine

IPD SHARING:
Plan to Share IPD: No
Any additional information regarding individual participants is available from the principle investigator of this study upon reasonable request.